CLINICAL TRIAL: NCT01327820
Title: Study of Post-operative Oxygen Consumption Following Vascular Surgery
Status: Completed | Type: Observational
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2011/R/AN/01; 11/S1102/1 (Other: South East Scotland Research Ethics Committee)
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Oxygen Consumption; Aortic Aneurysm; Peripheral Arterial Disease
Keywords: Oxygen consumption; Aortic Aneurysm; Peripheral Arterial Disease
MeSH Terms: conditions — Aortic Aneurysm; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Open aortic aneurysm repair
- Endovascular aortic aneurysm repair
- Infra-inguinal lower limb revascularisation

SUMMARY:
To define any changes in whole body oxygen consumption that occur following major vascular surgery (open aortic aneurysm surgery; endovascular aortic aneurysm repair; and infra-inguinal lower limb revascularisation procedures).

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for major vascular surgery at the Royal Infirmary of Edinburgh

Exclusion Criteria:

* Patient refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting for major vascular surgery at the Royal Infirmary of Edinburgh
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Whole body oxygen consumption | post-operative day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom